CLINICAL TRIAL: NCT03564691
Title: A Phase 1 Open Label, Multi-Arm, Multicenter Study of MK-4830 as Monotherapy and in Combination With Pembrolizumab for Participants With Advanced Solid Tumors
Brief Title: Study of MK-4830 as Monotherapy and in Combination With Pembrolizumab (MK-3475) in Participants With Advanced Solid Tumors (MK-4830-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4830-001; MK-4830-001 (Other: MSD); 2023-509542-35-00 (Registry Identifier: EU CT); U1111-1300-1952 (Registry Identifier: UTN); 2019-003164-53 (EudraCT Number)
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Neoplasms
Keywords: PD1; PD-1; PDL1; PD-L1
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab; Carboplatin; Pemetrexed; lenvatinib; Paclitaxel; Taxes; Cisplatin

STUDY DESIGN:
Intervention Model Description: Arms are parallel, except that participants who progress by either clinical or radiographic evaluation on monotherapy with MK-4830 (Dose Escalation, Part B), may switch over into the combination therapy arm of MK-4830 and pembrolizumab (Dose Escalation, Part C), provided they meet eligibility criteria. All arms are non-randomized except Dose Expansion Arms E and F, with randomization of eligible participants between those two arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (17):
- Dose Escalation, Part A: MK-4830 Monotherapy (Experimental): MK-4830 monotherapy (with MK-4830 doses determined by an accelerated titration design [ATD]) will be administered intravenously (IV), every 3 weeks (Q3W), starting with Cycle 1, Day 1, for a maximum of 35 cycles (up to approximately 2 years). Each cycle is 21 days. Participants enroll with histologically or cytologically confirmed pancreatic adenocarcinoma.
  Interventions: Drug: MK-4830
- Dose Escalation, Part B: MK-4830 Monotherapy (Experimental): MK-4830 monotherapy (with MK 4830 doses determined by a modified toxicity probability interval [mTPI] method) will be administered IV, Q3W, starting with Cycle 1, Day 1, for a maximum of 35 cycles (up to approximately 2 years). Each cycle is 21 days. Participants enroll with histologically or cytologically confirmed pleural or peritoneal malignant mesothelioma, epithelial, sarcomatoid, or biphasic subtypes.
  Interventions: Drug: MK-4830
- Dose Escalation, Part C: MK-4830 and Pembrolizumab (Experimental): Combination therapy with MK-4830 and pembrolizumab (with MK-4830 doses determined by an mTPI design). MK-4830 will be administered IV following pembrolizumab infusion, Q3W, starting with Cycle 1, Day 1, for a maximum of 35 cycles. Each cycle is 21 days. Pembrolizumab will be administered by IV, Q3W, starting with Cycle 1, Day 1. Each cycle is 21 days. The combination may be administered for a maximum of 35 cycles (up to approximately 2 years).
  Interventions: Drug: MK-4830; Drug: Pembrolizumab
- Dose Expansion, Arm A: Pancreatic Adenocarcinoma (Experimental): Combination therapy with the preliminary recommended phase 2 dose (RP2D) A of MK-4830, and pembrolizumab, in participants with histologically or cytologically confirmed pancreatic adenocarcinoma. MK-4830 will be administered IV following pembrolizumab infusion, Q3W, starting with Cycle 1, Day 1, for a maximum of 35 cycles. Each cycle is 21 days. Pembrolizumab will be administered by IV, Q3W, starting with Cycle 1, Day 1. Each cycle is 21 days. The combination may be administered for a maximum of 35 cycles (up to approximately 2 years).
  Interventions: Drug: MK-4830; Drug: Pembrolizumab
- Dose Expansion, Arm B: Glioblastoma (GBM) (Experimental): Combination therapy with the preliminary RP2D A of MK-4830, and pembrolizumab, in participants with histologically or cytologically confirmed GBM. MK-4830 will be administered IV following pembrolizumab infusion, Q3W, starting with Cycle 1, Day 1, for a maximum of 35 cycles. Each cycle is 21 days. Pembrolizumab will be administered by IV, Q3W, starting with Cycle 1, Day 1. Each cycle is 21 days. The combination may be administered for a maximum of 35 cycles (up to approximately 2 years).
  Interventions: Drug: MK-4830; Drug: Pembrolizumab
- Dose Expansion, Arm C: R/M HNSCC (Experimental): Combination therapy with the preliminary RP2D A of MK-4830, and pembrolizumab, in participants who have histologically or cytologically-confirmed recurrent or metastatic head and neck squamous cell carcinoma (R/M HNSCC) whose disease progressed on an anti-programmed cell death 1/programmed cell death ligand 1 (PD1/L1) therapy. MK-4830 will be administered IV following pembrolizumab infusion, Q3W, starting with Cycle 1, Day 1, for a maximum of 35 cycles. Each cycle is 21 days. Pembrolizumab will be administered by IV, Q3W, starting with Cycle 1, Day 1. Each cycle is 21 days. The combination may be administered for a maximum of 35 cycles (up to approximately 2 years).
  Interventions: Drug: MK-4830; Drug: Pembrolizumab
- Dose Expansion, Arm D: PD-L1 positive HNSCC, Dose A (Experimental): Combination therapy with the preliminary RP2D A of MK-4830, and pembrolizumab, in participants who have histologically or cytologically-confirmed advanced programmed death-ligand 1 (PD-L1) positive head and neck squamous cell carcinoma (HNSCC). MK-4830 will be administered IV following pembrolizumab infusion, Q3W, starting with Cycle 1, Day 1, for a maximum of 35 cycles. Each cycle is 21 days. Pembrolizumab will be administered by IV, Q3W, starting with Cycle 1, Day 1. Each cycle is 21 days. The combination may be administered for a maximum of 35 cycles (up to approximately 2 years).
  Interventions: Drug: MK-4830; Drug: Pembrolizumab
- Dose Expansion, Arm E: First-Line Advanced NSCLC, Dose A (Experimental): Combination therapy with the preliminary RP2D A of MK-4830, and pembrolizumab, in participants who have histologically-confirmed, first-line treatment advanced non-small-cell-lung-cancer (NSCLC) (Stage IIIB or IV). MK-4830 will be administered IV following pembrolizumab infusion, Q3W, starting with Cycle 1, Day 1, for a maximum of 35 cycles. Each cycle is 21 days. Pembrolizumab will be administered by IV, Q3W, starting with Cycle 1, Day 1. Each cycle is 21 days. The combination may be administered for a maximum of 35 cycles (up to approximately 2 years).
  Interventions: Drug: MK-4830; Drug: Pembrolizumab
- Dose Expansion, Arm F: First-Line Advanced NSCLC, Dose B (Experimental): Combination therapy with the preliminary RP2D B of MK-4830, and pembrolizumab, in participants who have histologically-confirmed, first-line treatment advanced non-small-cell-lung-cancer (NSCLC) (Stage IIIB or IV). MK-4830 will be administered IV following pembrolizumab infusion, Q3W, starting with Cycle 1, Day 1, for a maximum of 35 cycles. Each cycle is 21 days. Pembrolizumab will be administered by IV, Q3W, starting with Cycle 1, Day 1. Each cycle is 21 days. The combination may be administered for a maximum of 35 cycles (up to approximately 2 years).
  Interventions: Drug: MK-4830; Drug: Pembrolizumab
- Dose Expansion, Arm G: NSCLC, +Carboplatin/Pemetrexed (Experimental): Combination therapy with the preliminary RP2D A of MK-4830, pembrolizumab, and carboplatin/pemetrexed in participants with advanced non-squamous non-small-cell-lung-cancer (NSCLC) (Stage IIIB or IV). MK-4830 will be administered IV following pembrolizumab infusion, Q3W, starting with Cycle 1, Day 1, for a maximum of 35 cycles. Each cycle is 21 days. Pembrolizumab will be administered by IV, Q3W, starting with Cycle 1, Day 1. Each cycle is 21 days. The combination may be administered for a maximum of 35 cycles. Carboplatin and pemetrexed will be administered IV Q3W, starting with Cycle 1, Day 1, for 4 cycles, followed by pemetrexed Q3W continuous with MK-4830 and pembrolizumab, up to 35 cycles. Each cycle is 21 days (up to approximately 2 years).
  Interventions: Drug: MK-4830; Drug: Pembrolizumab; Drug: Carboplatin; Drug: Pemetrexed
- Dose Expansion, Arm H: RCC, +Lenvatinib (Experimental): Combination therapy with the preliminary RP2D A of MK-4830, pembrolizumab, and lenvatinib in participants with advanced renal cell carcinoma (RCC). MK-4830 will be administered IV, Q3W, starting with Cycle 1 following pembrolizumab infusion, Day 1, for a maximum of 35 cycles. Each cycle is 21 days. Pembrolizumab will be administered by IV, Q3W, starting with Cycle 1, Day 1. Each cycle is 21 days. The combination may be administered for a maximum of 35 cycles (up to approximately 2 years). Lenvatinib will be administered orally once daily for up to 35 cycles of 21 days (up to approximately 2 years).
  Interventions: Drug: MK-4830; Drug: Pembrolizumab; Drug: Lenvatinib
- Dose Expansion, Arm I: R/M Gastric/GE Junction Adenocarcinoma (Experimental): Combination therapy with the preliminary RP2D A of MK-4830, and pembrolizumab, in participants who have histologically or cytologically-confirmed recurrent or metastatic (R/M) gastric or gastroesophageal (GE) junction adenocarcinoma and who have been previously treated with at least 2 prior lines of therapy. MK-4830 will be administered IV following pembrolizumab infusion, Q3W, starting with Cycle 1, Day 1, for a maximum of 35 cycles. Each cycle is 21 days. Pembrolizumab will be administered by IV, Q3W, starting with Cycle 1, Day 1. Each cycle is 21 days. The combination may be administered for a maximum of 35 cycles (up to approximately 2 years).
  Interventions: Drug: MK-4830; Drug: Pembrolizumab
- Dose Expansion, Arm J: Ovarian Cancer (Experimental): Triple combination therapy with pembrolizumab plus preliminary RP2D A of MK-4830 plus paclitaxel in participants who have histologically confirmed, ovarian cancer. MK-4830 will be administered IV following pembrolizumab infusion, Q3W, starting with Cycle 1, Day 1, for a maximum of 35 cycles. Each cycle is 21 days. Pembrolizumab will be administered by IV, Q3W, starting with Cycle 1, Day 1 for a maximum of 35 cycles (up to approximately 2 years). Each cycle is 21 days. Paclitaxel will be administered by IV, once every week (QW) on Days 1, 8, and 15 of each 21-day cycle until disease progression or prohibitive toxicity.
  Interventions: Drug: MK-4830; Drug: Pembrolizumab; Drug: Paclitaxel
- Dose Expansion, Arm K: Triple negative Breast Cancer (TNBC) (Experimental): Triple combination therapy with pembrolizumab plus preliminary RP2D A of MK-4830 plus paclitaxel in participants who have histologically confirmed TNBC. MK-4830 will be administered IV following pembrolizumab infusion, Q3W, starting with Cycle 1, Day 1, for a maximum of 35 cycles. Each cycle is 21 days. Pembrolizumab will be administered by IV, Q3W, starting with Cycle 1, Day 1 for a maximum of 35 cycles (up to approximately 2 years). Each cycle is 21 days. Paclitaxel will be administered by IV on Days 1, 8, and 15 every 4 weeks (Q4W) until disease progression or prohibitive toxicity.
  Interventions: Drug: MK-4830; Drug: Pembrolizumab; Drug: Paclitaxel
- Dose Expansion, Arm L: Mesothelioma (Experimental): Triple combination therapy with pembrolizumab plus preliminary RP2D A of MK-4830 plus pemetrexed plus cisplatin in participants who have histologically confirmed advanced mesothelioma. MK-4830 will be administered IV following pembrolizumab infusion, Q3W, starting with Cycle 1, Day 1, for a maximum of 35 cycles. Each cycle is 21 days. Pembrolizumab will be administered by IV, Q3W, starting with Cycle 1, Day 1 for a maximum of 35 cycles (up to approximately 2 years). Each cycle is 21 days. Pemetrexed will be administered by IV, on Day 1 of each Q3W cycle for a maximum of 6 cycles. Each cycle is 21 days. Cisplatin will be administered by IV, on Day 1 of each Q3W cycle for a maximum of 6 cycles. Each cycle is 21 days.
  Interventions: Drug: MK-4830; Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Cisplatin
- Dose Expansion, Arm M: Advanced Solid Tumor in Chinese Participants In China (Experimental): Combination therapy with the preliminary RP2D A of MK-4830, and pembrolizumab, in Chinese participants, who reside in China, have histologically or cytologically-confirmed advanced/metastatic solid tumor, and who have been previously treated with at least 2 prior lines of therapy. MK-4830 will be administered IV following pembrolizumab infusion, Q3W, starting with Cycle 1, Day 1, for a maximum of 35 cycles. Each cycle is 21 days. Pembrolizumab will be administered by IV, Q3W, starting with Cycle 1, Day 1. Each cycle is 21 days. The combination may be administered for a maximum of 35 cycles (up to approximately 2 years).
  Interventions: Drug: MK-4830; Drug: Pembrolizumab
- Coformulation Phase, Arm N: MK-4830A (Coformulation of MK-4830 + pembrolizumab) (Experimental): Monotherapy with MK-4830A, a coformulation of MK-4830 800 mg + pembrolizumab 200 mg, in participants with histologically or cytologically-confirmed advanced/metastatic solid tumor, and who and have received, been intolerant to, been ineligible for, or refused all treatment known to confer clinical benefit. MK-4830A will be administered IV, Q3W, starting with Cycle 1, Day 1, for a maximum of 35 cycles (up to approximately 2 years). Each cycle is 21 days.
  Interventions: Biological: MK-4830A

INTERVENTIONS:
Drug: MK-4830 — MK-4830 will be administered intravenously (IV) Q3W. In Part C, MK-4830 will be administered after completion of pembrolizumab infusion. Dose escalation will proceed based on emerging safety and tolerability data of MK-4830 as monotherapy (Part A and B) and as combination therapy with pembrolizumab (Part C). For each dose level, an assessment will be made of the safety and tolerability data in order to define the next dose level to be tested.
  Arms: Dose Escalation, Part A: MK-4830 Monotherapy; Dose Escalation, Part B: MK-4830 Monotherapy; Dose Escalation, Part C: MK-4830 and Pembrolizumab; Dose Expansion, Arm A: Pancreatic Adenocarcinoma; Dose Expansion, Arm B: Glioblastoma (GBM); Dose Expansion, Arm C: R/M HNSCC; Dose Expansion, Arm D: PD-L1 positive HNSCC, Dose A; Dose Expansion, Arm E: First-Line Advanced NSCLC, Dose A; Dose Expansion, Arm F: First-Line Advanced NSCLC, Dose B; Dose Expansion, Arm G: NSCLC, +Carboplatin/Pemetrexed; Dose Expansion, Arm H: RCC, +Lenvatinib; Dose Expansion, Arm I: R/M Gastric/GE Junction Adenocarcinoma; Dose Expansion, Arm J: Ovarian Cancer; Dose Expansion, Arm K: Triple negative Breast Cancer (TNBC); Dose Expansion, Arm L: Mesothelioma; Dose Expansion, Arm M: Advanced Solid Tumor in Chinese Participants In China
Drug: Pembrolizumab — Pembrolizumab will be administered at 200 mg IV Q3W.
  Other Names: MK-3475; SCH 900475; KEYTRUDA®
  Arms: Dose Escalation, Part C: MK-4830 and Pembrolizumab; Dose Expansion, Arm A: Pancreatic Adenocarcinoma; Dose Expansion, Arm B: Glioblastoma (GBM); Dose Expansion, Arm C: R/M HNSCC; Dose Expansion, Arm D: PD-L1 positive HNSCC, Dose A; Dose Expansion, Arm E: First-Line Advanced NSCLC, Dose A; Dose Expansion, Arm F: First-Line Advanced NSCLC, Dose B; Dose Expansion, Arm G: NSCLC, +Carboplatin/Pemetrexed; Dose Expansion, Arm H: RCC, +Lenvatinib; Dose Expansion, Arm I: R/M Gastric/GE Junction Adenocarcinoma; Dose Expansion, Arm J: Ovarian Cancer; Dose Expansion, Arm K: Triple negative Breast Cancer (TNBC); Dose Expansion, Arm L: Mesothelioma; Dose Expansion, Arm M: Advanced Solid Tumor in Chinese Participants In China
Drug: Carboplatin — Carboplatin will be administered IV Q3W.
  Other Names: Paraplatin
  Arms: Dose Expansion, Arm G: NSCLC, +Carboplatin/Pemetrexed
Drug: Pemetrexed — Pemetrexed will be administered IV Q3W.
  Other Names: ALIMTA®; Pleumet; Pemecad
  Arms: Dose Expansion, Arm G: NSCLC, +Carboplatin/Pemetrexed; Dose Expansion, Arm L: Mesothelioma
Drug: Lenvatinib — Lenvatinib will be administered orally once daily.
  Other Names: LENVIMA®; Lenvanix
  Arms: Dose Expansion, Arm H: RCC, +Lenvatinib
Drug: Paclitaxel — Paclitaxel will be administered IV QW on Days 1, 8, and 15 of each 21-day cycle until disease progression or prohibitive toxicity (Arm J) and on Days 1, 8, and 15 Q4W until disease progression or prohibitive toxicity (Arm K).
  Other Names: Nov-Onxol; Onxol; Paclitaxel Novaplus; Taxol
  Arms: Dose Expansion, Arm J: Ovarian Cancer; Dose Expansion, Arm K: Triple negative Breast Cancer (TNBC)
Drug: Cisplatin — Cisplatin will be administered IV Q3W.
  Other Names: Platinol®; Platinol®-AQ; CDDP
  Arms: Dose Expansion, Arm L: Mesothelioma
Biological: MK-4830A — MK-4830A, a coformulation of MK-4830 800 mg + pembrolizumab 200 mg, will be administered IV Q3W.
  Arms: Coformulation Phase, Arm N: MK-4830A (Coformulation of MK-4830 + pembrolizumab)

SUMMARY:
This study consists of several parts: dose escalation, dose expansion, dose expansion in Chinese participants residing in China, and coformulation. Dose escalation is to evaluate the safety, tolerability, and preliminary efficacy of MK-4830 monotherapy administration (Arms A and B) and in combination with pembrolizumab (Arm C). Dose expansion is to evaluate the objective response rate (ORR) of MK-4830 in combination with pembrolizumab (Arms A-F); evaluate the safety and tolerability of MK-4830 administered in combination with pembrolizumab, carboplatin, and pemetrexed (Arm G) and of MK-4830 administered in combination with pembrolizumab and lenvatinib (Arm H); evaluate the safety, tolerability and ORR of MK-4830 in combination with pembrolizumab plus chemotherapy (Arms I-L); and evaluate the safety and tolerability of MK-4830 in combination with pembrolizumab in Chinese participants from China (Arm M). The coformulation part (Arm N) evaluates the safety and tolerability of MK-4830A (coformulation of MK-4830 800 mg + pembrolizumab 200 mg). There is no formal hypothesis testing in this study.

ELIGIBILITY:
Inclusion Criteria:

* Dose escalation participants: Has any histologically- or cytologically-confirmed advanced/metastatic solid tumor by pathology report and has received, has been intolerant to, or has been ineligible for all treatment known to confer clinical benefit. Solid tumors of any type are eligible for enrollment
* Has measurable disease by Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1), Response Assessment in Neuro-Oncology (RANO), or modified RECIST (mRECIST) as assessed by the local site investigator/radiology
* Submits an evaluable baseline tumor sample for analysis (either a recent or archival tumor sample). This inclusion criterion does not apply to Expansion phase Arm M
* Dose Escalation Part C and Back-fill participants: Has 1 or more discrete malignant lesions that are amenable to biopsy
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale. This inclusion criterion does not apply to Expansion phase Arm B
* Demonstrates adequate organ function
* A male participant must agree to use an approved contraception(s) during the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm during this period
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and either not a woman of childbearing potential (WOCBP) OR if a WOCBP agrees to follow the study contraceptive guidance during the treatment period and for at least 180 days after the last dose of study treatment
* Expansion phase Arm A participants:

  * Has histologically or cytologically confirmed metastatic pancreatic adenocarcinoma
  * Received at least 1 prior line of therapy and no more than 3 prior lines of systemic therapy
* Expansion phase Arm B participants:

  * Has histologically or cytologically confirmed unresectable glioblastoma multiforme (GBM) or its variants
  * Has a Karnofsky performance status (KPS) ≥ 70
  * Has had no more than 1 prior line of therapy for GBM. Radiation with or without chemotherapy is acceptable as the prior treatment
  * Has shown unequivocal evidence for tumor progression by magnetic resonance imaging (MRI) or computed tomography (CT) scan by contrast within 2 weeks prior to randomization
  * Has an interval of at least 3 weeks (to randomization) between prior surgical resection (one week for stereotactic biopsy)
  * Has an interval of at least 12 weeks from the completion of radiation therapy to randomization unless there is unequivocal histologic confirmation of tumor progression or radiographic progression outside of the prior radiation field
  * Is neurologically stable (eg, without a progression of neurologic symptoms or requiring escalating doses of systemic steroid therapy within last 2 weeks) and clinically stable
* Expansion phase Arm C participants:

  * Has histologically confirmed recurrent or metastatic head and neck squamous cell cancer (HNSCC) of the oral cavity, oropharynx, hypopharynx, and/or larynx that is considered incurable by local therapies
  * Has experienced disease progression at any time during or after treatment with a platinum-containing (eg, carboplatin or cisplatin) regimen with or without cetuximab
* Expansion phase Arm D participants:

  * Has histologically confirmed advanced or metastatic HNSCC of the oral cavity, oropharynx, hypopharynx, and/or larynx that is considered incurable by local therapies
  * Has not had any prior programmed cell death 1 (PD-1)/ programmed cell death ligand 1 (PD-L1) therapy
* Expansion phase Arms E and F participants:

  * Has a histologically or cytologically confirmed diagnosis of advanced (Stage IIIb) or Stage IV metastatic non-small-cell lung cancer (NSCLC)
  * Has received no prior systemic therapy for chemotherapy or other targeted or biological antineoplastic therapy treatment for Stage IIIb or Stage IV metastatic NSCLC. Treatment with chemotherapy and/or radiation as part of neoadjuvant/adjuvant therapy is allowed if therapy was completed at least 6 months prior to the diagnosis of advanced disease. Participants with prior treatment with an anti-PD-1 or PD-L1 agent are not eligible
* Expansion phase Arm G participants:

  * Has a histologically or cytologically confirmed diagnosis of advanced (Stage IIIb) or Stage IV metastatic nonsquamous NSCLC (American Joint Committee on Cancer (AJCC) version 8)
  * Is able to tolerate chemotherapy with carboplatin and pemetrexed
  * Has received no prior systemic therapy for advanced NSCLC
* Expansion phase Arm H participants:

  * Has histologically confirmed diagnosis of renal cell cancer (RCC) with clear cell component with or without sarcomatoid features
  * Has locally advanced/metastatic disease or has recurrent disease
  * May have received 1 or 2 prior lines of systemic therapy for advanced RCC
* Expansion phase Arm I participants:

  * Has histologically confirmed diagnosis of recurrent and/or metastatic gastric or gastroesophageal junction adenocarcinoma that is considered incurable by local therapies
  * Has received and progressed on at least two prior chemotherapy regimens
  * If tumor was if human epidermal growth factor receptor 2 (HER2/neu) positive, participant must have previously received treatment with trastuzumab
* Expansion phase Arm J participants

  * Has histologically confirmed high-grade epithelial ovarian, fallopian tube or primary peritoneal carcinoma
  * Has received 1 or 2 prior lines of systemic therapy, including at least 1 prior platinum-based therapy
  * Has radiographic evidence of disease progression
  * Is a candidate for paclitaxel chemotherapy
* Expansion phase Arm K participants:

  * Has locally recurrent inoperable breast cancer OR have metastatic breast cancer not previously treated
  * Has confirmed triple-negative breast cancer (TNBC)
  * Has completed treatment for Stage I-III breast cancer, if indicated, and ≥6 months elapsed between the completion of treatment and first documented local or distant disease recurrence
  * Has been treated with (neo)adjuvant anthracycline
* Expansion phase Arm L participants:

  * Has histologically confirmed diagnosis of recurrent and/or advanced mesothelioma that is considered incurable by standard therapies
  * Is eligible to receive standard chemotherapy
* Expansion phase Arm M participants

  * Has any histologically or cytologically confirmed advanced/metastatic solid tumor by pathology report and have received, been intolerant of, been ineligible for, or refused all treatment known to confer clinical benefit
  * Has received up to 2 prior systemic regimens for the treatment of advanced/metastatic solid tumor
  * Is a Chinese participant residing in China
* Coformulation Arm N participants

  * Has any histologically- or cytologically-confirmed advanced/metastatic solid tumor by pathology report and have received, been intolerant to, been ineligible for, or refused all treatment known to confer clinical benefit

Exclusion Criteria:

* Has had chemotherapy, definitive radiation, or biological cancer therapy within 4 weeks (2 weeks for palliative radiation) prior to the first dose of study therapy, or has not recovered from any adverse events (AEs) that were due to cancer therapeutics administered more than 4 weeks earlier
* Has not recovered from all radiation-related toxicities to Grade 1 or less, requires corticosteroids, and had radiation pneumonitis
* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years
* Has known untreated central nervous system metastases or known carcinomatous meningitis. This exclusion criterion does not apply to Expansion phase Arm B
* Has received any prior immunotherapy and was discontinued from that treatment due to a Grade 3 or higher immune-related AEs
* Has previously had a severe hypersensitivity reaction to treatment with a monoclonal antibody or has a known sensitivity to any component of pembrolizumab and/or chemotherapy agents
* Has an active infection requiring therapy
* Has a history or current interstitial lung disease
* Has a history of noninfectious pneumonitis that required steroids or current pneumonitis
* Has an active autoimmune disease that has required systemic treatment in the past 2 years except vitiligo or resolved childhood asthma/atopy
* Has clinically significant cardiac disease, including unstable angina, acute myocardial infarction within 6 months from Day 1 of study drug administration, or New York Heart Association Class III or IV congestive heart failure
* Has a known history of human immunodeficiency virus (HIV)
* Has a known active hepatitis B or C
* Is taking chronic systemic steroids in doses >10 mg daily of prednisone or equivalent within 7 days prior to the first dose of trial treatment
* Has not fully recovered from any effects of major surgery without significant detectable infection. Surgical proceduress that required general anesthesia must be completed at least 2 weeks before first study treatment administration. Surgery requiring regional/epidural anesthesia must be completed at least 72 hours before first study treatment administration and participants should be recovered
* Has received a live or live-attenuated virus vaccine within 30 days prior to first dose of study intervention
* Is currently participating and receiving study therapy in a study of an investigational agent or has participated and received study therapy in a study of an investigational agent or has used an investigational device within 28 days of administration of MK-4830
* All Expansion phase participants:

  * Tumor types with known MSI-high status are not eligible
* Expansion phase Arm A participants:

  * Has received more than 3 lines of prior therapy for advanced disease (pancreatic cancer)
* Expansion phase Arm B participants:

  * Has tumor primarily localized to the brainstem or spinal cord
  * Has presence of diffuse leptomeningeal disease or extracranial disease
  * Has recurrent tumor greater than 6 cm in maximum diameter
  * Requires treatment with moderate or high dose systemic corticosteroids for at least 3 days within 2 weeks of randomization
* Expansion phase Arm D participants:

  * Has received prior systemic chemotherapy or other targeted or biological antineoplastic therapy treatment for their advanced metastatic HNSCC
* Expansion phase Arm E and F participants:

  * Has received prior systemic chemotherapy or other targeted or biological antineoplastic therapy treatment for their Stage IIIb or Stage IV metastatic NSCLC
  * Has had prior treatment with any anti-PD-1, PD-L1, or programmed cell death-ligand 2 (PD-L2) agent
* Expansion phase Arm G participants:

  * Has received prior systemic chemotherapy or other targeted or biological antineoplastic therapy treatment for their Stage IIIb or Stage IV nonsquamous NSCLC
  * Has had prior treatment with any anti-PD-1, PD-L1, or PD-L2 agent
* Expansion phase Arm H participants:

  * Has a clinically significant gastrointestinal (GI) abnormality
  * Has a history of untreated deep vein thrombosis or pulmonary embolism within 6 months prior to screening
  * Has poorly controlled hypertension
  * Has active GI bleeding
  * Has evidence of inadequate wound healing
  * Has active bleeding disorder or other history of significant bleeding episodes within 30 days prior to randomization
  * Has hemoptysis within 6 weeks prior to randomization
  * Has radiographic evidence of encasement or invasion of a major blood vessel, or of intratumoral cavitation
* Expansion phase Arm I participants:

  * Has experienced weight loss > 10 % over 2 months prior to first dose of study therapy
  * Has clinical evidence of ascites
  * Has peritoneal metastases
* Expansion phase Arm J participants:

  * Has non-epithelial cancers, including borderline, malignant Müllerian mixed mucinous, malignant Brenner's tumor and undifferentiated carcinoma and/or germ cell tumors and/or sex cord - stromal tumors
  * Has received more than 2 prior lines of systemic therapy for ovarian cancer
* Expansion phase Arm K participants:

  * Has a known history of hypersensitivity or allergy to the study chemotherapies and/or any of their components
* Expansion phase Arm L participants:

  * Has a known history of hypersensitivity or allergy to the study chemotherapies and/or any of their components
  * Is receiving any medication prohibited in combination with study chemotherapies as described in the respective product labels, unless medication was stopped within 7 days prior to randomization
* All Participants (Arms A through N)

  * Has symptomatic pleural effusion (eg, cough, dyspnea, pleuritic chest pain)
  * Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicities (DLTs) | Cycle 1 (Up to 21 days)
  The occurrence of the following toxicities, if assessed by the investigator to be possibly, probably, or definitely related to study treatment administration:
  * Grade 4 nonhematologic toxicity (not laboratory)
  * Grade 4 hematologic toxicity lasting >=7 days, except thrombocytopenia:
  * Any nonhematologic AE >=Grade 3 in severity, with exceptions
  * Any Grade 3 or Grade 4 alanine aminotransferase, aspartate aminotransferase, and/or bilirubin laboratory value
  * Any other nonhematologic laboratory value if:
  Clinically significant medical intervention is required to treat the participant, OR The abnormality leads to hospitalization, OR The abnormality persists for >1 week, OR The abnormality results in a drug-induced liver injury
  * Febrile neutropenia Grade 3 or Grade 4
  * Prolonged delay (>2 weeks) in initiating Cycle 2 due to treatment-related toxicity.
  * Any treatment-related toxicity that causes the participant to discontinue treatment during Cycle 1.
  * Grade 5 toxicity
Number of Participants Who Experienced an Adverse Event (AE) | Up to approximately 27 months
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. The number of participants who experienced an AE will be presented.
Number of Participants Who Discontinued Study Treatment Due to an AE | Up to approximately 24 months
  An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. The number of participants who discontinued study treatment due to an AE will be presented.
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or Response Assessment in Neuro-Oncology (RANO) as Assessed by Investigator | Up to approximately 24 months
  For Arms A, C-F, I, and K ORR is defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. For Arm B, ORR is defined as the percentage of participants who experience a PR or CR per RANO, determined by: disappearance or size reduction of lesions, and review of abnormalities on fluid-attenuated inversion recovery (T2/FLAIR) images; Clinical status based on age-adjusted performance; And whether daily steroid dose has changed since previous visit. The percentage of participants who experience a CR or PR based on modified RECIST 1.1 as assessed by investigator or based on RANO will be presented.
ORR per Modified RECIST (mRECIST) 1.1 as Assessed by Investigator | Up to approximately 24 months
  Per protocol, ORR per mRECIST 1.1 will be reported for Arm L participants. ORR is defined as percentage of participants who have CR (disappearance of all pleural & non-pleural disease) or PR (summed measurement (SM) decrease by at least 30% from baseline scan SM) per mRECIST 1.1. The percentage of participants who experience CR or PR based on mRECIST 1.1 as assessed by investigator will be presented.

SECONDARY OUTCOMES:
Area Under the Curve (AUC) of Plasma MK-4830 | At designated time points detailed in Description (Up to approximately 25 months)
  Pharmacokinetic (PK) parameter: area under the drug concentration/time curve. Samples will be drawn 24 hours pre-MK-4830 infusion and end of infusion on Day 1 of Cycles 1, 2, 4, 6, and 8, and every 4 cycles thereafter (plus cycle 3 for Dose Expansion Arms) and 2 hours post-infusion on Day 1 of Cycles 1, 2, 4, 6, and 8 (plus cycle 3 for Dose Expansion Arms); on Days 8 and 15 for cycle 1, and additionally in cycles 2-3 for Dose Escalation Arms only; and at time of drug Discontinuation and 30 days after last dose (Up to approximately 25 months). Dose Expansion Arm C additionally requires the above pre-, post-, and 2 hour post-dose samples on Day 3 of Cycle 1. Each cycle is 21 days.
Minimum Concentration Between Doses (Ctrough) of Plasma MK-4830 | At designated time points detailed in Description (Up to approximately 25 months)
  PK parameter: minimum drug concentration between doses. Samples will be drawn 24 hours pre-MK-4830 infusion and end of infusion on Day 1 of Cycles 1, 2, 4, 6, and 8, and every 4 cycles thereafter (plus cycle 3 for Dose Expansion Arms) and 2 hours post-infusion on Day 1 of Cycles 1, 2, 4, 6, and 8 (plus cycle 3 for Dose Expansion Arms); on Days 8 and 15 for cycle 1, and additionally in cycles 2-3 for Dose Escalation Arms only; and at time of drug Discontinuation and 30 days after last dose (Up to approximately 25 months). Dose Expansion Arm C additionally requires the above pre-, post-, and 2 hour post-dose samples on Day 3 of Cycle 1. Each cycle is 21 days.
Maximum Drug Concentration (Cmax) of Plasma MK-4830 | At designated time points detailed in Description (Up to approximately 25 months)
  PK parameter: maximum drug concentration. Samples will be drawn 24 hours pre-MK-4830 infusion and end of infusion on Day 1 of Cycles 1, 2, 4, 6, and 8, and every 4 cycles thereafter (plus cycle 3 for Dose Expansion Arms) and 2 hours post-infusion on Day 1 of Cycles 1, 2, 4, 6, and 8 (plus cycle 3 for Dose Expansion Arms); on Days 8 and 15 for cycle 1, and additionally in cycles 2-3 for Dose Escalation Arms only; and at time of drug Discontinuation and 30 days after last dose (Up to approximately 25 months). Dose Expansion Arm C additionally requires the above pre-, post-, and 2 hour post-dose samples on Day 3 of Cycle 1. Each cycle is 21 days.
Number of Participants Positive for Anti-Drug Antibodies (ADA) After MK-4830 plus Pembrolizumab Treatment | At designated time points (Up to approximately 25 months)
  Serum samples from participants treated with MK-4830 plus pembrolizumab will be analyzed for ADA using a neutralizing antibody assay. The number of participants positive for ADA will be reported.
Minimum Concentration Between Doses (Ctrough) of Plasma Pembrolizumab in Arm M | At designated time points detailed in Description (Up to approximately 25 months)
  PK parameter: minimum drug concentration between doses. Samples will be drawn 24 hours pre-pembrolizumab infusion on Day 1 of Cycles 1-4, 6, 8, and every 4 cycles thereafter; post-infusion on Day 1 of Cycle 1; and at time of drug Discontinuation and 30 days after last dose (Up to approximately 25 months). Each cycle is 21 days.
Maximum Drug Concentration (Cmax) of Plasma Pembrolizumab in Arm M | At designated time points detailed in Description (Up to approximately 25 months)
  PK parameter: maximum drug concentration. Samples will be drawn 24 hours pre-pembrolizumab infusion on Day 1 of Cycles 1-4, 6, 8, and every 4 cycles thereafter; post-infusion on Day 1 of Cycle 1; and at time of drug Discontinuation and 30 days after last dose (Up to approximately 25 months). Each cycle is 21 days.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (37):
- United States (9):
  - University of California at San Francisco ( Site 0004), San Francisco, California
  - Henry Ford Health System ( Site 0002), Detroit, Michigan
  - Washington University ( Site 0003), St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0005), Hackensack, New Jersey
  - Laura and Isaac Perlmutter Cancer Center ( Site 0008), New York, New York
  - Ohio State University Arthur G James Cancer Hospital & Richard J Solove Research Institute ( Site 00, Columbus, Ohio
  - South Texas Accelerated Research Therapeutics, LLC (START) ( Site 0001), San Antonio, Texas
  - Utah Cancer Specialists ( Site 0011), Salt Lake City, Utah
  - Seattle Cancer Care Alliance ( Site 0010), Seattle, Washington
- Australia (2):
  - Liverpool Hospital-Medical Oncology ( Site 0250), Liverpool, New South Wales
  - Princess Alexandra Hospital ( Site 0253), Brisbane, Queensland
- Canada (3):
  - Juravinski Cancer Centre ( Site 0034), Hamilton, Ontario
  - The Ottawa Hospital ( Site 0031), Ottawa, Ontario
  - Princess Margaret Cancer Centre ( Site 0033), Toronto, Ontario
- China (3):
  - The First Hospital of Jilin University ( Site 0803), Changchun, Jilin
  - Shanghai Chest Hospital-Oncology department ( Site 0801), Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University ( Site 0804), Chengdu, Sichuan
- France (3):
  - Centre Oscar Lambret ( Site 2002), Lille, Nord
  - Centre Hospitalier Universitaire de Poitiers ( Site 2000), Poitiers, Vienne
  - Hôpital Européen Georges Pompidou ( Site 2003), Paris, Île-de-France Region
- Greece (3):
  - University General Hospital of Heraklion ( Site 0110), Heraklion, Irakleio
  - Euromedica General Clinic of Thessaloniki-Oncology Unit ( Site 0112), Thessaloniki
  - European Interbalkan Medical Center ( Site 0111), Thessaloniki
- Israel (4):
  - Rambam Health Care Campus-Oncology Division ( Site 0042), Haifa
  - Rabin Medical Center ( Site 0043), Petah Tikva
  - Chaim Sheba Medical Center. ( Site 0044), Ramat Gan
  - Sourasky Medical Center ( Site 0041), Tel Aviv
- Japan (2):
  - National Cancer Center Hospital East ( Site 0400), Kashiwa, Chiba
  - Japanese Foundation for Cancer Research ( Site 0401), Tokyo
- Poland (2):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie (, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne ( Site 0151), Gdansk, Pomeranian Voivodeship
- South Africa (3):
  - Wits Clinical Research ( Site 0213), Johannesburg, Gauteng
  - The Oncology Centre ( Site 0212), Durban, KwaZulu-Natal
  - Cancercare Rondebosch Oncology ( Site 0210), Cape Town, Western Cape
- Severance Hospital Yonsei University Health System ( Site 0300), Seoul, South Korea
- Spain (2):
  - Instituto Catalan de Oncologia ICO - Hospital Duran i Reynals ( Site 0101), L'Hospitalet de Llobregat, Barcelona
  - Centro Integral Oncologico Clara Campal START Madrid ( Site 0102), Madrid

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Siu LL, Wang D, Hilton J, Geva R, Rasco D, Perets R, Abraham AK, Wilson DC, Markensohn JF, Lunceford J, Suttner L, Siddiqi S, Altura RA, Maurice-Dror C. First-in-Class Anti-immunoglobulin-like Transcript 4 Myeloid-Specific Antibody MK-4830 Abrogates a PD-1 Resistance Mechanism in Patients with Advanced Solid Tumors. Clin Cancer Res. 2022 Jan 1;28(1):57-70. doi: 10.1158/1078-0432.CCR-21-2160. Epub 2021 Oct 1. PMID 34598945
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26332&tenant=MT_MSD_9011